CLINICAL TRIAL: NCT02233985
Title: A Randomized Trial of Nebulized 3% Hypertonic Saline With Salbutamol in the Treatment of Acute Bronchiolitis in Pediatric Hospital
Brief Title: Nebulized 3% Hypertonic Saline Solution Treatment of Bronchiolitis in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-2012-1002-43
Record Dates: First submitted 2014-05-07; First posted 2014-09-09 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2012-12

CONDITIONS: Bronchiolitis; Wheezing
Keywords: bronchiolitis; hypertonic; saline; salbutamol
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebulized 0.9% Sodium Chloride (Active Comparator): Salbutamol 100 micrograms / kg / dose administered 0.9 % saline solution (4ml) nebulized for 3 initial sessions lasting 20 minutes each and every 4 hours during the entire hospital stay.
  Interventions: Drug: 0.9% Sodium Chloride
- Nebulized 3% Sodium Chloride (Experimental): Salbutamol 100 micrograms / kg / dose administered 3 % saline solution (4ml) nebulized for 3 initial sessions lasting 20 minutes each and every 4 hours during the entire hospital stay.
  Interventions: Drug: 3% Sodium Chloride

INTERVENTIONS:
Drug: 0.9% Sodium Chloride — Salbutamol 100 micrograms / kg / dose administered 0.9% saline solution (4ml) nebulized for 3 initial sessions lasting 20 minutes each and every 4 hours during the entire hospital stay.
  Other Names: 0.9% saline
  Arms: Nebulized 0.9% Sodium Chloride
Drug: 3% Sodium Chloride — Salbutamol 100 micrograms / kg / dose administered 3 % saline solution (4ml) nebulized for 3 initial sessions lasting 20 minutes each and every 4 hours during the entire hospital stay.
  Other Names: 3% saline
  Arms: Nebulized 3% Sodium Chloride

SUMMARY:
- Determine the efficacy of nebulized salbutamol/hypertonic saline combination in moderate to severe bronchiolitis.

DETAILED DESCRIPTION:
* Study design: double-blind, randomized, parallel-controlled prospective study.
* Location: Department of pediatric emergencies and pediatric hospitalization of Highly Specialized Medical Unit (HSMU), Hospital of Gynecology-Obstetrics and Paediatrics (HGOP) No. 48, Mexican Institute of Social Security (MISS).
* Patients: 50 patients were included; 25 for each group. Patients had between 2 and 24 months of age with a first episode of wheezing associated with respiratory distress and a history of infection of the upper respiratory tract, with moderate to severe degree of respiratory distress according to the Respiratory Distress Scale of Sant Joan de Déu Hospital (SJDH) .
* Interventions: the randomly allocated patients received in group I nebulised 0.9% saline with salbutamol 100 micrograms / kg / dose for 3 initial sessions lasting 20 minutes each and every 4 hours. In group II , hypertonic (3%) saline plus salbutamol 100 micrograms / kg / dose for 3 initial sessions lasting 20 minutes each and every 4 hours. In both groups, will be performed at baseline Scale SJDH Respiratory Distress and the end of the first 3 sessions, you will have 30 minutes to make the second evaluation and at 4 hours the third at 8 hours and then every 24 hours throughout the hospital stay . The independent variable is the intervention with hypertonic saline 3% and the variable primary outcome will be assessed improvement or cure with Respiratory Distress Scale SJDH and secondary outcome will be the time of hospital stay .
* Descriptive statistics of all variables will be reported. T test was used for two independent groups or nonparametric test according to the distribution of the variables to compare the clinical improvement between the groups with the Scale of Respiratory Distress SJDH, as well as to determine whether there is a difference in time of hospital stay between the two study groups. Square test or Fisher exact chi used to compare readmissions for bronchial hyperresponsiveness between the two groups as well as the complications of the disease itself in each study group. Be reported with frequencies and percentages side effects of hypertonic saline 3%. Was considered statistically significant p <0.05. The results with the Number Cruncher Statistical System (NCSS) 2004 statistical program will be discussed.
* The sample size was calculated with t-test to compare means of continuous variables, resulting in 25 subjects per group.
* In the follow-up period it was possible to obtain more patients from the baseline estimate of the sample number.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients aged 2 months to 24 months of age, both genders attending the pediatric emergency service.
* With first episode of wheezing associated with respiratory distress and a history of upper respiratory tract infection.
* You have the evaluation of respiratory difficulty with Scale Hospital Sant Joan de Deu (HSJD) from 6 to 16 at entry points (moderate and severe degree).

Exclusion Criteria:

* Subjects with a history of previous wheezing, asthma, or who have received bronchodilator treatment before the present illness.
* Subjects with chronic lung disease, with heart disease, with congenital or acquired anatomic abnormalities of the airway.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-08; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria P Sosa-Bustamante, MD, Study Director — Unidad Medica de Alta Especialidad Bajio 48. Hospital de Gineco - Pediatria. Instituto Mexicano del Seguro Social
Locations (1):
- Unidad Medica de Alta Especialidad Bajío No. 48 Hospital de Gineco - Pediatría. Instituto Mexicano del Seguro Social, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
We have your membership number social security and personal data such as address and telephone number of the parents.

REFERENCES:
- [Background] Kuzik BA, Flavin MP, Kent S, Zielinski D, Kwan CW, Adeleye A, Vegsund BC, Rossi C. Effect of inhaled hypertonic saline on hospital admission rate in children with viral bronchiolitis: a randomized trial. CJEM. 2010 Nov;12(6):477-84. doi: 10.1017/s1481803500012690. PMID 21073773
- [Background] Sharma BS, Gupta MK, Rafik SP. Hypertonic (3%) saline vs 0.93% saline nebulization for acute viral bronchiolitis: a randomized controlled trial. Indian Pediatr. 2013 Aug;50(8):743-7. doi: 10.1007/s13312-013-0216-8. Epub 2012 Dec 5. PMID 23502662
- [Background] Gupta N, Puliyel A, Manchanda A, Puliyel J. Nebulized hypertonic-saline vs epinephrine for bronchiolitis; proof of concept study of cumulative sum (CUSUM) analysis. Indian Pediatr. 2012 Jul;49(7):543-7. doi: 10.1007/s13312-012-0122-5. Epub 2010 Oct 30. PMID 22080619
- [Background] Al-Ansari K, Sakran M, Davidson BL, El Sayyed R, Mahjoub H, Ibrahim K. Nebulized 5% or 3% hypertonic or 0.9% saline for treating acute bronchiolitis in infants. J Pediatr. 2010 Oct;157(4):630-4, 634.e1. doi: 10.1016/j.jpeds.2010.04.074. Epub 2010 Jun 19. PMID 20646715
- [Background] Luo Z, Fu Z, Liu E, Xu X, Fu X, Peng D, Liu Y, Li S, Zeng F, Yang X. Nebulized hypertonic saline treatment in hospitalized children with moderate to severe viral bronchiolitis. Clin Microbiol Infect. 2011 Dec;17(12):1829-33. doi: 10.1111/j.1469-0691.2010.03304.x. Epub 2010 Jul 15. PMID 20636429
- [Background] Grewal S, Ali S, McConnell DW, Vandermeer B, Klassen TP. A randomized trial of nebulized 3% hypertonic saline with epinephrine in the treatment of acute bronchiolitis in the emergency department. Arch Pediatr Adolesc Med. 2009 Nov;163(11):1007-12. doi: 10.1001/archpediatrics.2009.196. PMID 19884591
- [Background] Luo Z, Liu E, Luo J, Li S, Zeng F, Yang X, Fu Z. Nebulized hypertonic saline/salbutamol solution treatment in hospitalized children with mild to moderate bronchiolitis. Pediatr Int. 2010 Apr;52(2):199-202. doi: 10.1111/j.1442-200X.2009.02941.x. Epub 2009 Aug 7. PMID 19674354
- [Background] Postiaux G, Louis J, Labasse HC, Gerroldt J, Kotik AC, Lemuhot A, Patte C. Evaluation of an alternative chest physiotherapy method in infants with respiratory syncytial virus bronchiolitis. Respir Care. 2011 Jul;56(7):989-94. doi: 10.4187/respcare.00721. Epub 2011 Feb 22. PMID 21352671

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebulized 0.9% Sodium Chloride | Nebulized 3% Sodium Chloride
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In the follow-up period it was possible to obtain more patients from the baseline estimate of the sample number.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized 0.9% Sodium Chloride | Nebulized 3% Sodium Chloride | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.7 (5.7) | 8.8 (5.7) | 8.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 16 | 20 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 31 | 64
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Score Respiratory Distress
Description: It is a validated clinical scale, sufficiently reliable measure of Severity of the respiratory distress. It consists of the summation score of the sibilance / crackling parameters (the largest of them), respiratory effort, pulmonary air inlet, oxygen saturation, heart rate and breathing rate. It is stratified into 3 levels of severity: mild from 0 to 5 points, moderate from 6 to 10 and severe from 10 to 16.
Time Frame: Basal, 30 minutes after the end of the first 3 continuous nebulization sessions, at 4 hours, 8 hours and every 24 hours during the entire hospital stay
Population: All patients with respiratory distress in moderate to severe stage until a stage of mild respiratory distress or difficulty breathing submitted.
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- Hypertonic Saline Solution 3% (HSS 3%) Group; Saline Solution 0.9% (SS 0.9%) Group: Patients with moderate stages (6 to 10 points) and severe (11 to 16 points) were selected, performing subsequent measurements always 30 minutes after nebulization corresponding.
Arm/Group | Hypertonic Saline Solution 3% (HSS 3%) Group | Saline Solution 0.9% (SS 0.9%) Group
Number analyzed (Participants) | 31 | 33
units on a scale
  Basal | 8 [7 to 10] | 8 [8 to 10]
  30 minutes | 6 [5 to 7] | 8 [8 to 9]
  4 hours | 5 [3 to 6] | 8 [7 to 9]
  8 hours | 3 [3 to 5] | 8 [6 to 9]
  12 hours | 3 [2 to 7] | 7 [6 to 9]
  24 hours | 0 [0 to 0] | 7 [6 to 9]
  48 hours | 0 [0 to 0] | 7 [6 to 9]
  72 hours | 0 [0 to 0] | 6 [3 to 7]
  96 hours | 0 [0 to 0] | 5 [4 to 9]
  120 hours | 0 [0 to 0] | 3 [3 to 3]
  144 hours | 0 [0 to 0] | 6 [6 to 6]
  196 hours | 0 [0 to 0] | 4 [4 to 4]

2. Primary Outcome: Hours of Hospital Stay
Description: Each patient record the time of entry and measured the total hospital stay time in hours, recording the time of discharge to determine the total stay in hours. The hospital stay will be evaluated in hours. Staying hospitalized until they had mild respiratory stage scale scores for at least 2 hrs.
Time Frame: Throughout the stay for each patient until discharge. Follow-up will be continued for a period of 30 days in which they may present readmissions, complications or adverse effects.
Population: All patients included in the study, underwent measurement of hours of hospital stay from admission to pediatric emergencies to hospital discharge.
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Hypertonic Saline Solution 3% (SHS 3%); Saline Solution 0.9% (SS 0.9%) Group: We counted the hours from admission of the patient to the pediatric emergency department until hospital discharge. Staying hospitalized until they had mild respiratory stage scale scores for at least 2 hrs.
Arm/Group | Hypertonic Saline Solution 3% (SHS 3%) | Saline Solution 0.9% (SS 0.9%) Group
Number analyzed (Participants) | 31 | 33
hours | 8 [5.4 to 9] | 39.3 [23.9 to 61.6]

3. Secondary Outcome: Hospital Readmission
Description: After the first admission of each patient will be evaluated during the next 30 days, if a patient is readmitted for any respiratory disease, respiratory distress, pneumonia or bronchiolitis. Considering as non-serious risks that do not compromise life, tachycardia, tremor, increased access to cough immediately to the inhalation, as well as the ardor of nasal mucosa, all these with limited characteristics, however, these do not put at risk The health of the patient, so they were not measured.
Time Frame: as for outcome 2
Reporting Status: Not Posted, anticipated posting 2017-05

4. Secondary Outcome: Frequency of Complications of the Disease Itself
Description: The presence or absence of clinical data to warrant dehydration of hydration, infected by bacteria, pneumothorax, interstitial emphysema and subcutaneous be evaluated.
Time Frame: as for outcome 2
Reporting Status: Not Posted, anticipated posting 2017-05

ADVERSE EVENTS:
Time Frame: 1 month
Description: Since their admission to the trial, until a month after discharge.
Arm/Group | Nebulized 0.9% Sodium Chloride | Nebulized 3% Sodium Chloride
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No